CLINICAL TRIAL: NCT07201909
Title: Can A Prebiotic Fibre bLend Improve Stress, Mood, and Anxiety? Assessing the Impact of a Daily Prebiotic Fibre Blend on Affect, Inflammation, and the Gut Microbiome: a 12-week Double-blind Placebo-controlled RCT
Brief Title: CALM Study: Can A Prebiotic Fibre bLend Improve Stress, Mood, and Anxiety?
Acronym: CALM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Myota GmbH (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CALM
Record Dates: First submitted 2025-08-14; First posted 2025-10-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Stress
Keywords: gut-brain axis; perceived stress; prebiotic fibre; cognitive function; anxiety; mood; depression; inflammation
MeSH Terms: conditions — Anxiety Disorders; Depression; Inflammation

STUDY DESIGN:
Intervention Model Description: Two-arm, double-blind, placebo-controlled randomised trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic fibre blend (Experimental): Prebiotic fibre blend, consisting of 10g of a powdered supplement, to be taken daily alongside usual diet for 12 weeks.
  Interventions: Dietary Supplement: Prebiotic fibre blend
- Placebo (Placebo Comparator): Placebo will be 10g of maltodextrin powder, to be taken daily alongside usual diet for 12 weeks.
  Interventions: Dietary Supplement: Maltodextrin powder

INTERVENTIONS:
Dietary Supplement: Prebiotic fibre blend — A blend of prebiotic fibres in a powdered supplement form.
  Arms: Prebiotic fibre blend
Dietary Supplement: Maltodextrin powder — Maltodextrin powder
  Arms: Placebo

SUMMARY:
This clinical trial will investigate whether a powdered prebiotic fibre blend can improve perceived stress levels in healthy adults with mild-moderate stress levels.

DETAILED DESCRIPTION:
There is growing interest in how the gut microbiota interacts with the brain to influence psychological outcomes, particularly stress. Even in otherwise healthy individuals, persistent psychological stress is associated with measurable physiological changes-including elevated cortisol levels, heightened hypothalamic-pituitary-adrenal (HPA) axis reactivity, and systemic low-grade inflammation. These biological signatures are increasingly understood to be shaped, in part, by the composition and activity of the gut microbiota.

In this study, we're investigating how a powdered prebiotic fibre supplement can improve stress levels. You may have heard people refer to this as the 'gut-brain axis'. We'll also be looking at the link between the prebiotic fibre supplement intake and changes in other areas of health, like depression, mood, anxiety, cognition, inflammation, and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years of age
* Capacity to give informed consent to participate in the study
* Able to comply with study requirements and visits
* Meet the range required for mild-moderate stress levels (as assessed by DASS-42 stress subscale)
* Normal or corrected to normal vision and/or hearing

Exclusion Criteria:

* Current smoker
* Having food allergies and/or intolerances
* Diagnosis of Type 1 or 2 diabetes or cardiovascular disease or psychiatric or neurological conditions (e.g. schizophrenia, dementia) including eating disorders
* Current or previous diagnosis of depression in past 6 months
* Receiving medications that lower cholesterol, blood pressure, blood glucose levels, or improve insulin sensitivity
* Receiving antidepressant or anti-anxiety medications or treatments
* Receiving hormonal birth control
* Perimenopause or menopause
* Pregnancy, lactation, or an intent to become pregnant during the course of the study
* Continuous antibiotic use for > 3 days within 1 month prior to enrolment
* Continuous use of weight-loss drug for > 1 month before screening
* Major change in dietary intake in past month (e.g. excluding whole food groups)
* Currently consuming daily prebiotic or probiotic supplements
* Prior use (< 6 months) of any blood glucose or cholesterol lowering medication
* Any significant GI condition affecting GI absorption including (but not limited to) inflammatory bowel disease, weight loss surgery, irritable bowel disease.
* End stage renal disease
* Active cancer, or treatment for any cancer, in last 3 years
* Consuming more than 20g of fibre a day as assessed by the 18-item FiberScreen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | Baseline and 12 weeks
  The primary objective is to determine the effect of 12-week long daily administration of Prebiotic fibre blend as compared to Placebo on stress scores (Perceived Stress Scale) on a scale between 0 - 40 (where higher scores indicate higher stress).

SECONDARY OUTCOMES:
Perceived Stress | Baseline and 8 weeks
  To determine the effect of 12-week long daily administration of Prebiotic fibre blend as compared to Placebo on stress scores (Perceived Stress Scale) on a scale between 0 - 40 (where higher scores indicate higher stress).
Depression | Baseline, 8 weeks, and 12 weeks
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on depression scores (DASS-42), on a scale between 0 - 21 (where higher scores mean higher depression).
Mood | Baseline, 8 weeks and 12 weeks
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on mood scores (PANAS-X), on a scale between 10 - 50 (where higher scores on the Positive Affect scale indicate higher levels of positive engagement with your environment; while higher scores on the Negative Affect scale indicate higher levels of negative engagement).
Anxiety | Baseline, Week 8, and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on anxiety scores (DASS-42), on a scale between 0 - 21 (where higher scores mean higher anxiety levels).
Serum hs-CRP | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on serum high sensitivity C-Reactive Protein (hs-CRP).
Gastrointestinal symptoms | Baseline, Week 8, and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on gastrointestinal symptoms (GSRS), on a scale of 15 - 105 where higher scores indicate more severe gastrointestinal discomfort.
Cognition: Emotional Stroop | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on emotional interference in attention and processing (reaction time and accuracy), as assessed by the Emotional Stroop where better scores are achieved by lower reaction times and higher accuracy score.
Cognition: Affective 2-Back Task | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on emotional interference in working memory under emotional load, as assessed by the Affective 2-Back Task, where better scores are achieved by lower reaction times and higher accuracy score.
Cognition: Emotional Go-No-Go | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on emotion-related inhibitory control and response suppression, as assessed by the Emotional Go-No-Go, where better scores are achieved by higher correct response rates and lower commission errors.
Cognition: Number-Letter Task | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on cognitive flexibility and task-switching ability, as assessed by the Number-Letter Task, where better scores are achieved by higher numbers of correctly recalled items.
Cognition: Attentional Network Task | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on efficiency of alerting, orienting, and executive attention networks, as assessed by the Attentional Network Task , where better scores are achieved by lower reaction times and higher accuracy.

OTHER OUTCOMES:
Sleep Quality | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on sleep quality (PSQI), on a scale of 0 - 21 where higher scores indicate worse sleep.
Quality of Life Index | Baseline And Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on quality of life index (WHOQOL), on a scale of 0 -100 where higher scores indicate higher quality of life.
Serum LDL Cholesterol | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on serum LDL cholesterol.
Serum HDL Cholesterol | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on serum HDL cholesterol.
Serum Triglycerides | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on serum triglycerides.
Total cholesterol | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on serum total cholesterol.
Waist to hip ratio | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on waist to hip ratio.
Waist circumference | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on waist circumference (cm).
Gut microbiome composition | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on gut microbiome diversity scores (alpha and beta measures) and composition (differential abundance testing).
Systolic blood pressure | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on systolic blood pressure (mmHg).
Diastolic blood pressure | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on diastolic blood pressure (mmHg).
BMI | Baseline and Week 12
  To determine the effect of 12-week daily administration of Prebiotic fibre blend as compared to Placebo on BMI (kg/m2).
Exploratory endpoint | Baseline, Week 8, and Week 12
  Inter-dependencies between primary and secondary outcomes will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- CALM Study Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared.